CLINICAL TRIAL: NCT00137826
Title: Phase II Study of Bevacizumab (Avastin) and Erlotinib (Tarceva) in Previously Treated Malignant Mesothelioma
Brief Title: Bevacizumab (Avastin) and Erlotinib (Tarceva) in Previously Treated Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Pasi A. Janne, MD, PhD, Associate Professor, Medicine, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-369
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Mesothelioma
Keywords: Mesothelioma; Avastin; Bevacizumab; Tarceva; OSI-774; Erlotinib
MeSH Terms: conditions — Mesothelioma | interventions — Erlotinib Hydrochloride; Bevacizumab

INTERVENTIONS:
Drug: Erlotinib — Taken orally once daily. Participants may continue on study treatment until disease progresses or they experience serious side effects.
  Other Names: Tarceva; OSI-774
Drug: Bevacizumab — Given intravenously over 30-90 minutes, on day 1 of each 21-day cycle. Participants may continue on study treatment until disease progresses or they experience serious side effects.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine whether the combination of the investigational drugs Avastin and Tarceva are effective in patients with mesothelioma who have previously been treated with chemotherapy.

DETAILED DESCRIPTION:
Each cycle of study treatment lasts 21 days. The patient will take erlotinib by mouth once daily. On day 1 of every cycle, the patient will receive bevacizumab intravenously over a 30-90 minute time period.

CT scan(s), MRI(s) and/or x-ray(s) of the cancer site will be performed every 6 weeks (2 cycles) to assess the extent of the response to treatment.

Bloodwork will be performed before the first dose of erlotinib and bevacizumab at Cycle 1, Cycle 2, Cycle 3, and at the end of treatment.

At the completion of the treatment a physical exam, vital signs, blood tests, urine tests and standard radiologic testing will be performed.

The duration of study depends upon how the patients' mesothelioma responds to treatment as well as how well the patient tolerates the medication.

ELIGIBILITY:
Inclusion Criteria:

* Mesothelioma that has been previously treated with at least one chemotherapy regimen
* 18 years of age or older
* Must at least be able to walk and capable of taking care of oneself although unable to carry out work activities
* Four or more weeks since last major surgery
* Four or more weeks since last radiation therapy
* Three or more weeks since last chemotherapy
* Life expectancy of 12 weeks or more
* Blood tests that show kidneys, liver and bone marrow to be working adequately
* Able to comply with study and/or follow-up procedures

Exclusion Criteria:

* Prior exposure to Tarceva (OSI-774, erlotinib), trastuzumab, ZD1839 or C225
* Receiving anticoagulation medication other than low dose Coumadin
* Clinically significant heart disease such as uncontrolled hypertension, previous heart attack within past 12 months, uneven heartbeat, etc.
* History of central nervous system disease such as seizures not controlled with standard medical therapy, brain metastases or history of stroke
* Major surgery within 28 days of screening
* Daily treatment with aspirin or anti-inflammatory medications
* Pregnant or lactating (pertaining to women only)
* Serious or nonhealing wound, ulcer or bone fracture
* Difficulty swallowing
* A disease or disorder that interferes with ability to digest and absorb food
* History of coughing up more than 1/4 teaspoon of blood
* A medical condition that could make it unsafe for patient to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the response to the combination of bevacizumab and erlotinib in previously treated malignant mesothelioma | 3 years

SECONDARY OUTCOMES:
To determine the time to tumor progression
to determine the duration of response
to determine the median and overall survival of patients
to determine the safety of the drugs administered | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Janne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - The University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Perez-Soler R, Chachoua A, Hammond LA, Rowinsky EK, Huberman M, Karp D, Rigas J, Clark GM, Santabarbara P, Bonomi P. Determinants of tumor response and survival with erlotinib in patients with non--small-cell lung cancer. J Clin Oncol. 2004 Aug 15;22(16):3238-47. doi: 10.1200/JCO.2004.11.057. PMID 15310767
- See also: Dana-Farber Cancer Institute Lowe Thoracic Oncology Program — http://www.dana-farber.org/Adult-Care/Treatment-and-Support/Lung-Cancer,-Non-Small-Cell.aspx